CLINICAL TRIAL: NCT05639374
Title: Effectiveness of a Peer-led Program to Prevent Alcohol Consumption. A Randomized Controlled Trial.
Brief Title: Effectiveness of a Peer-led Program to Prevent Alcohol Consumption.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Asociación de Amigos, Universidad de Navarra (Unknown); Banco Santander (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CODIGO
Record Dates: First submitted 2022-11-24; First posted 2022-12-06 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Drinking
Keywords: Peer; Alcohol drinking; Health promotion; Undergraduate; Brief Motivational Intervention
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BASICS_HealthyClassroom (Experimental): Students assigned to the IG will receive the peer-led preventive program. The preventive program consists of a single face-to-face session, lasting about 45-50 minutes. First, the participant will receive, from the Research Staff in Training, the individualized feedback sheet prepared from the baseline information obtained through the "BASICS_HealthyClassroom Questionnaire". Subsequently, they will have a motivational interview with the counsellor. The content of the intervention will be adapted to the interests and level of motivation of each participant.
  Interventions: Behavioral: BASICS_HealthyClassroom
- Control Group (No Intervention): Students assigned to the CG will not receive any type of intervention, they will only receive the usual information and messages that students receive in their daily environments and at the University.

INTERVENTIONS:
Behavioral: BASICS_HealthyClassroom — First, they will complete a 22-item online questionnaire, collecting all the variables of the research. After completing it, the students in the intervention group will receive personalized feedback by mail that visually summarizes the content of the questionnaire. Students will receive a motivational intervention with the aim of increasing the university's awareness of their alcohol consumption. In the intervention session of the program, the following aspects may be addressed, whenever the participant wishes: 1) Pattern of alcohol consumption of the student; 2) Social norm of alcohol consumption; 3) Negative consequences of alcohol; 4) Costs of alcohol consumption; 5) The change; 6) Specific education on alcohol; and 7) Advice and recommendations.
  Arms: BASICS_HealthyClassroom

SUMMARY:
The goal of this Randomized clinical trial is to evaluate the effectiveness of a peer-led intervention to prevent alcohol consumption in university students. The main questions it aims to answer are:

* Does a peer-led brief motivational intervention reduce the quantity and frequency of alcohol consumption among university students?
* Does a peer-led brief motivational intervention reduce the negative consequences experienced by university students due to alcohol consumption?

Participants will:

* Complete a baseline online questionnaire (before the intervention) and one month after receiving the intervention.
* Participants in the intervention group will receive a brief motivational intervention.

Researchers will compare intervention and control group to see if there are statistically significant differences in relation to alcohol consumption.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary Objectives:

1. To evaluate the effectiveness of a peer-led program to prevent alcohol consumption in university students.
2. To compare the effectiveness of said program with a control group that will obtain the usual information and messages that students receive in their daily environments and at the University.

Secondary objectives:

1. Evaluate the acquisition by the peer counsellors of the micro-skills of motivational interviewing (MI).
2. Evaluate the adherence of peer counsellors to the content of the program to prevent excessive alcohol consumption.
3. To explore the experience of peer counsellors when carrying out the alcohol consumption prevention intervention with their peers.

Program objectives:

1. Decrease the amount of alcohol consumed in a normal week and weekend in students receiving the intervention compared to those in the control group.
2. Reduce episodes of binge drinking in university students who receive the intervention program.
3. Reduce estimated peak blood alcohol concentration (eBAC) in students receiving the intervention program.
4. Reduce the number of negative consequences experienced by the students derived from alcohol consumption.

Hypothesis:

1. An educational program, with an emphasis on improving motivation and empowerment, and led by trained peer counsellors, will be more effective in preventing the harmful use of alcohol in university students than the usual health promotion that this population receives.
2. Students in the intervention group will decrease the amount of alcohol consumed in a normal week and weekend compared to those in the control group, and this difference between the two groups will be clinically relevant.
3. The students who receive the intervention will experience fewer episodes of binge drinking compared to the university students in the control group.
4. Students in the intervention group will reduce the estimated peak blood alcohol concentration compared to those in the control group.
5. Students in the intervention group will experience fewer negative consequences from alcohol use compared to those in the control group.
6. Students receiving the intervention will be more motivated to make positive changes in their alcohol risk behaviour compared to the control group.

STUDY METHODOLOGY

Sample and setting:

In the Randomized Clinical Trial, 306 university students will be randomized to two treatment groups: intervention (IG) and control (CG). The research will be carried out from September 2022 to May 2023 at the University of Navarra (Pamplona). The study population will be made up of first-year university students of the Degree in Nursing, Sciences, Pharmacy and Nutrition, Communication, Law, Economics and Business, Education and Psychology, and Philosophy of a university in the north of Spain, enrolled in the academic year 2022/ 2023.

Study procedure:

The study participants will complete the "BASICS_HealthyClassroom Questionnaire" which is carried out through the "Survey Monkey" platform. This is self-completed in a time of 15 minutes, consists of a total of 22 questions.

Student volunteers who complete the baseline survey and who meet the inclusion criteria will be randomized to one of the two treatment conditions (IG or CG) and will subsequently be contacted by mail to inform them of their selection in the project. Students assigned to the intervention group will receive the peer-led preventive program. The preventive program consists of a single face-to-face session, lasting about 45-50 minutes. In the first place, the participant will receive, from the Research Staff in Training, the individualized feedback sheet prepared from the baseline information obtained through the "BASICS_HealthyClassroom Questionnaire". Later, they will have a motivational interview with the peer counselor (approximately 45 minutes). The content of the intervention will be adapted to the interests and level of motivation of each participant.

The data will be collected in three times. Before the intervention (Time 0; T0), and one month after the intervention (T1).

The peer counselors who carry out the intervention will be fourth-year students from the Faculty of Nursing of the University, who will have previously been trained to carry out the intervention program. The training is being carried out in the first quarter of the 2022-2023 academic year, as part of the optional subject "Motivational Interviewing and Process of Change" of the Faculty of Nursing of the University of Navarra, offered to fourth-year students. . The subject consists of, on the one hand, theoretical classes given by an expert on the subject (10h) and, on the other hand, MI practice workshops and feedback (13h).

The effectiveness of the intervention will be evaluated through the change in the pattern of alcohol consumption, and the negative consequences experienced by each participant.

Recruitment will take place during the month of November (2022) through the transmission of direct information about the project in the first-year undergraduate classes at the faculties involved, and through dissemination on social networks and the website of the University.

The motivational interventions will take place from January to March, when the peer counselors have finished the training.

ELIGIBILITY:
Inclusion Criteria:

* University students who are in their first or second year of studies.
* Having had at least one episode of heavy alcohol consumption or binge drinking in the last month.
* Students with availability to attend the intervention.
* Students with mobile phone availability.
* Students who understand and can communicate well in Spanish.

Exclusion Criteria:

* Students who have repeated the course and it is not their first year at the University.
* Students who have previously studied another career.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline total number of alcoholic beverages consumed in a normal week and weekend (including Thursday, Friday and Saturday) at one month. | Baseline, T1 (one month)
  It will be measured by self-declaration of the participant using the modified version of the Daily Drinking Questionnaire. In this instrument the participant enters each day of the week the number of alcoholic beverages consumed. The greater the number of drinks, the greater the risk of alcohol consumption.
Change from Baseline frequency of binge drinking episodes (in the last month), at one month. | Baseline, T1 (one month)
  It will be measured by self-declaration of the participant using a specific closed question. In the case of men it will be: "Think about the last month. How many days have you had 5 or more glasses, pints or glasses of alcoholic beverages on the same occasion of consumption (for example, the same night)?"; and for women: "Think about the last month. How many days have you had 4 or more glasses, pints or glasses of alcoholic beverages on the same occasion of consumption (for example, the same night)? Participants answer the number of days they binge drink. The higher the number, the consumption is more risky.
Change from Baseline estimated peak alcohol concentration reached on the occasion of highest consumption, at one month. | Baseline, T1 (one month)
  It will be measured by self-declaration of the participant using the Quantity/Frequency/Peak Index.
  A self-report measure designed to assess a student's drinking behavior in terms of quantity and frequency of their alcohol consumption on a typical occasion and peak drinking occasion on a given occasion in the past month (number of alcoholic beverages ingested on the occasion of greatest consumption in the last month, and number of hours invested in their consumption). From this information, together with the participant's specific body weight and sex, a computer algorithm is used to estimate the normal and maximum blood alcohol concentration achieved. Blood alcohol levels are calculated as the ratio of milligrams of alcohol per 100 milliliters of blood, and are reported as a percentage.
  The higher the blood alcohol level, the more alcohol intoxication the participant will have suffered.
Change from Baseline short-term consequences of alcohol consumption, at one month. | Baseline, T1 (one month)
  It will be measured by self-declaration of the participant using the Spanish Version of the Young Adult Alcohol Consequences Questionnaire.
  It is an instrument that seeks to measure the negative consequences associated with alcohol consumption. This tool is made up of 48 items with a dichotomous response format (yes/no), through which the student must respond according to their experience during the last year. In this way, the total score ranges from 0 to 48, the higher the score, the greater the predisposition to develop problems and consequences related to the consumption of alcoholic beverages.

SECONDARY OUTCOMES:
Number of Motivational Interviewing micro-skills used by peer counsellors. | Right at the end of training, the last day of training.
  It will be collected through the observation and analysis of the intervention sessions, during the training, recorded on audio. The Peer Proficiency Assessment will be used.
  The tool allows obtaining a total score for each of the behaviors evaluated. Thus, for open and closed questions, the score is obtained by counting the number of questions observed. For simple and complex reflexes, one score is first obtained for each reflex subtype (i.e., repeat, rephrase, double-sided reflex, etc.) and then globally summed, thus obtaining two scores , one for simple reflexes and one for complex ones.
  In relation to the interpretation of the scores, the competence to carry out an effective peer counseling session is defined as the counselor-client interaction that meets a 1:1 ratio of open and closed questions, a 1:1 ratio of complex and simple reflections, and a 2:1 ratio of reflections to questions.
Number of topics addressed during the motivational interview. | Right at the end of training, the last day of training.
  It will be collected through the observation and analysis of the intervention sessions, during the training, recorded on audio. An ad-hoc checklist will be used.
  This tool consists of a list of statements regarding what the student should address during the intervention sessions, and which includes the theoretical content taught in the training of students on alcohol. When listening to the recording, the researcher marks with a cross those statements that have been made correctly.
  It consists of 27 topics, the greater the number of topics addressed, the more complete the motivational interview will have been.
Qualitative variable: Experience of the peer counselors when carrying out the motivational intervention with their peers. | Right at the end of training, the last day of training.
  It will be collected by self-declaration of the peer counselor through focus groups.

CONTACTS AND LOCATIONS:
Overall Officials: Navidad Canga Armayor, PhD, Principal Investigator — University of Navarra
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pilatti A, Read JP, Caneto F. Validation of the Spanish Version of the Young Adult Alcohol Consequences Questionnaire (S-YAACQ). Psychol Assess. 2016 May;28(5):e49-61. doi: 10.1037/pas0000140. Epub 2015 Aug 24. PMID 26302103
- [Background] Dimeff, L.A., Baer, J.S., Kivlahan, D.R., Marlatt, G.A. (1999). Brief Alcohol Screening and Intervention for College Students (BASICS): A Harm Reduction Approach. New York: Guilford Press.
- [Background] Mastroleo, N. R. (2008). Comparison of Supervision Training Techniques in a Motivational Enhancement Intervention on College Student Drinking [doctoral dissertation].The Pennsylvania State University.
- [Background] Collins RL, Parks GA, Marlatt GA. Social determinants of alcohol consumption: the effects of social interaction and model status on the self-administration of alcohol. J Consult Clin Psychol. 1985 Apr;53(2):189-200. doi: 10.1037//0022-006x.53.2.189. No abstract available. PMID 3998247
- [Derived] Lavilla-Gracia M, Pueyo-Garrigues M, Calavia Gil D, Esandi-Larramendi N, Alfaro-Diaz C, Canga-Armayor N. Peer-led BASICS intervention to reduce alcohol consumption and alcohol-related consequences among university students: a randomized controlled trial. Front Public Health. 2023 Oct 31;11:1280840. doi: 10.3389/fpubh.2023.1280840. eCollection 2023. PMID 38026297